CLINICAL TRIAL: NCT05773235
Title: MRI-markers to Monitor Small Vessel Disease Dynamics in the Prognosis of Small Vessel Disease-associated, Cerebrovascular Events - a Prospective Cohort Study
Brief Title: MRI-markers to Monitor Small Vessel Disease Dynamics in the Prognosis of Small Vessel Disease-associated, Cerebrovascular Events
Acronym: MRI-PRO-SVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02006
Record Dates: First submitted 2023-02-09; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Intracerebral Hemorrhage; CAA - Cerebral Amyloid Angiopathy; Cerebral Small Vessel Diseases
Keywords: Intracerebral hemorrhage; Ischemic stroke; Cerebral amyloid angiopathy; Hypertensive deep perforator arteriopathy; 7 Tesla-MRI; Cerebral small vessel disease; Ultra high-field MRI
MeSH Terms: conditions — Cerebral Hemorrhage; Cerebral Amyloid Angiopathy, Familial; Cerebral Small Vessel Diseases; Ischemic Stroke; Cerebral Amyloid Angiopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with intracerebral hemorrhage: Patients with symptomatic intracranial hemorrhage (defined as non-traumatic intracerebral hemorrhage or convexity, non-aneurysmal subarachnoid hemorrhage) enrolled in the PRO-SVD study
  Interventions: Diagnostic Test: Combined 3- and 7 Tesla-MRI
- Healthy controls: Clinically healthy persons of at least 55 years of age
  Interventions: Diagnostic Test: Combined 3- and 7 Tesla-MRI

INTERVENTIONS:
Diagnostic Test: Combined 3- and 7 Tesla-MRI — 7 Tesla-MRI including the following sequences: susceptibility weighted imaging (SWI), T1, T2, FLAIR, quantitative mapping sequences (T1mapping, qSM)

SUMMARY:
This is a nested cohort study in the PRO-SVD cohort. Small vessel disease is a chronic disease and is thought to progress over time. MRI is the gold standard to diagnose small vessel disease, but data on MRI-visible disease progression are scarce. Complications of small vessel disease as well as location pattern, distribution and severity of these MRI small vessel disease markers differ according to the underlying phenotype. The primary aim of this project is to investigate individual small vessel disease burden progression detected by MRI in survivors or intracerebral hemorrhage.

ELIGIBILITY:
For patients with intracerebral hemorrhage

Inclusion Criteria:

* Patient participating in the PRO-SVD cohort
* Symptomatic intracranial hemorrhage
* Written informed consent provided by patient or next-of-kin
* No contraindications against MRI

Exclusion Criteria:

* Patient unsuitable for MRI follow-ups (e.g. claustrophobia)
* Patients unlikely to attend 1-year follow-up

For healthy controls

Inclusion Criteria:

* Clinically healthy person ≥ 55 years
* Written informed consent provided by the healthy control
* No contraindications against MRI

Exclusion Criteria:

* Known or suspected cerebral small vessel diseases or presence of concurrent diseases potentially mimicking small vessel disease (e.g. multiple sclerosis, previous heart surgery etc.)
* Pre-existing dementia, cognitive decline or disorder of the central nervous system.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 consecutive patients with cerebral small vessel disease-related intracerebral hemorrhage admitted to the Inselspital Bern. Patients will undergo combined 3/7 Tesla-MRI according to a standardised small vessel disease MRI protocol at 3 timepoints.
  A control group consisting of 10 clinically asymptomatic subjects will undergo the same MRI protocol at one timepoint.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 24 months
  Composite endpoint of a new, clinically symptomatic ischaemic or haemorrhagic event as defined by the treating physician and/or any increase in small vessel disease and/or cerebral amyloid angiopathy burden according to small vessel disease burden score (range 0-4 points, higher score means higher small vessel disease burden) or cerebral amyloid angiopathy burden score (range 0-6 points, higher score means higher cerebral amyloid angiopathy burden), respectively.

SECONDARY OUTCOMES:
MRI-defined disease progression | 24 months
  Any increase in small vessel disease (SVD) and/or cerebral amyloid angiopathy (CAA) burden according to small vessel disease burden score (range 0-4 points, higher score means higher small vessel disease burden) or cerebral amyloid angiopathy burden score (range 0-6 points, higher score means higher cerebral amyloid angiopathy burden), respectively.
Increase in number of SVD-attributable, ischaemic lesions | 24 months
  Composite outcome defined as any increase in numeric count for lacunes and/or increase in perivascular space severity scale (0/1-10 PVS/11-20 PVS/21-40 PVS/>40 PVS) and/or increase in periventricular or deep separate white matter Fazekas scale.
Increase in number of SVD-attributable, haemorrhagic lesions | 24 months
  Composite outcome defined as any increase in numeric count for cerebral microbleeds and/or increase in cortical superficial siderosis multifocality score.
Increase in perivascular space severity scale | 24 months
  Defined as any increase in perivascular space (PVS) severity scale (0/1-10 PVS/11-20 PVS/21-40 PVS/>40 PVS, higher number of PVS means higher small vessel disease burden).
Clinical, vascular outcome event | 24 months
  Composite endpoint including any of the following, clinically apparent events:
  * ischaemic stroke as diagnosed by CT or MRI and causing a corresponding clinical deficit (as assessed by the treating physician)
  * intracerebral haemorrhage as diagnosed by CT or MRI and causing a corresponding clinical deficit (as assessed by the treating physician)
  * systemic vascular event defined as radiological or clinical evidence of arterial hypoperfusion and judged by the treating physician to be due to an atherosclerotic or embolic cause.
Functional outcome | 24 months
  Modified Rankin Scale (ordinal scale, range 0-6 with 0 corresponding to no symptoms at all and 6 corresponding to death).
New cognitive impairment | 24 months
  Montreal Cognitive Assessment (MoCA, range 0-30 points) < 26 points (corresponding to impaired cognitive function) and/or new impairment in activities of daily living as defined by the treating physician .

CONTACTS AND LOCATIONS:
Overall Officials: David J Seiffge, Prof, MD, Principal Investigator — Department of Neurology, Inselspital Bern University Hospital
Locations (1):
- Department of Neurology, Inselspital Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data sharing can be discussed by qualified researchers with the principal investigator upon reasonable request and might be subject to prior additional approval by the respective ethical board.